CLINICAL TRIAL: NCT02733861
Title: Evaluation of the Related Factors Influencing the Stability of Dental Implants
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Air Force Military Medical University, China (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Zhang Yumei, Professor, Air Force Military Medical University, China
Other Study IDs: IRB-REV-2016012
Record Dates: First submitted 2016-03-29; First posted 2016-04-12 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Teeth Missing
Keywords: dental implant; stability; implant stability quotient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
With the development of oral medicine,dental implants has become a very popular solution to remediate the loss of teeth and dental rehabilitation. For the last few decades, the immediate loading protocol have become more and more popular because the increasing demands of shortened treatment time. Implant stability is considered one of the most important parameters in implant dentistry. It affects the healing and successful osseointegration of implants. For any implant procedure, successful implant integration is a prerequisite criterion, which depends on a series of procedure-related and patient-dependent factors. It also has been considered that preoperative measurement is critical and may give valuable information to predict loading time and survival of the implants.

In this clinical study, the samples were collected from patients with single teeth missing who came from the department of prosthodontics from the School of Stomatology of the Fourth Military Medical University.The prospective cohort study was used to investigate the correlation between different factors and the early stability of the implants. And then, using the correlation between different factors and the early implant stability gives predictable data about implant stability and then evaluate the accuracy and reliability.

DETAILED DESCRIPTION:
Ethical and institutional approval was obtained from the study institution. From May 2015 to May 2017, teeth missing consecutive patients requiring implant treatment consented to participate in this study to investigate the correlation between implant stability and bone density.

Cone beam computed tomography (CBCT) was used for preoperative radiological evaluation of the jawbone for each patient, and then bone density in Houndsfield units scale was assessed by SimPlant Pro 11.04 software. Immediately after the implant placement and 12 weeks later, stability measurements were performed with Osstell™ Mentor.The captured data was represented in a quantitative unit called Implant Stability Quotient (ISQ) on a scale from 1 to 100 and averaged for each implant.

The descriptive statistical methods were used to show the differences in bone density and ISQ values among location, gender, age and implant diameter variables. Mann-whitney test was used for comparison of HU values and ISQ values between different age and gender groups. Kruskal-Wallis test was used for comparison of HU values and ISQ values between different location and implant diameter groups. The changes of ISQ values over time were compared using Wilcoxon signed rank test. The Spearman's rank correlation coefficient was used to investigate the correlation between ISQ values and HU values.

At last, to investigate the possible correlations between implant stability and bone density and to study the feasibility of predicting implant stability by using preoperative CBCT.

ELIGIBILITY:
Inclusion Criteria:

* the patients who had undergone tooth extraction within the previous 3 months

Exclusion Criteria:

* those who required bone augmentation simultaneously with implant insertion, and patients with any systemic disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: single teeth missing consecutive patients requiring implant treatment consented to participate in this study
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Implant stability quotient (ISQ) was tested by Osstell™ Mentor | on the day of surgery
  The transducer probe was aimed at the small magnet on top of the SmartPeg at a distance of 2 to 3 mm and held stable during the pulsing time until the instrument beeped and displayed the ISQ value. If two ISQ values were displayed simultaneously, their mean value was recorded. Measurements were taken twice in the buccolingual direction as well as in the mesiodistal direction. The mean of all measurements was rounded to the nearest whole number and was regarded as representative of the ISQ.
Implant stability quotient (ISQ) was tested by Osstell™ Mentor | on the 12th weeks after surgery
  The transducer probe was aimed at the small magnet on top of the SmartPeg at a distance of 2 to 3 mm and held stable during the pulsing time until the instrument beeped and displayed the ISQ value. If two ISQ values were displayed simultaneously, their mean value was recorded. Measurements were taken twice in the buccolingual direction as well as in the mesiodistal direction. The mean of all measurements was rounded to the nearest whole number and was regarded as representative of the ISQ.

SECONDARY OUTCOMES:
Measure the bone density of the implant locations by CBCT. | within 10 days before surgery
  Using the interactive setting on the SimplantTM software, an implant was then placed over the alveolar portion of each edentulous span to include the trabecular portion and the outer cortical shell when present. The computer was then asked to map the density of the bone around the entire circumference of each implant, with a surrounding thickness of 1 mm, which is the default setting . Multiple adjacent readings were taken within each span, where possible. Subsequently, all areas subjectively classified into each of the four qualities were pooled so that a range of Houndsfield values (HU) could be attributed to each particular quality, and a mean value was calculated in order to establish a new objective quantitative scale of bone density.
Measure the thickness of the bone around the implant by CBCT. | immediately after the surgery
  Using the interactive setting on the SimplantTM software, an implant was then placed over the alveolar portion of each edentulous span to include the trabecular portion and the outer cortical shell when present. The computer was then asked to map the density of the bone around the entire circumference of each implant, with a surrounding thickness of 1 mm, which is the default setting . Multiple adjacent readings were taken within each span, where possible. Subsequently, all areas subjectively classified into each of the four qualities were pooled so that a range of Houndsfield values (HU) could be attributed to each particular quality, and a mean value was calculated in order to establish a new objective quantitative scale of bone density.
Measure the crestal bone resorption by X-ray images | immediately and 3 months after the surgery
  The transducer probe was aimed at the small magnet on top of the SmartPeg at a distance of 2 to 3 mm and held stable during the pulsing time until the instrument beeped and displayed the ISQ value. If two ISQ values were displayed simultaneously, their mean value was recorded. Measurements were taken twice in the buccolingual direction as well as in the mesiodistal direction. The mean of all measurements was rounded to the nearest whole number and was regarded as representative of the ISQ.

CONTACTS AND LOCATIONS:
Overall Officials: Yumei Zhang, PhD, Principal Investigator — Department of prosthetic dentistry, Stomatology hospital, Fourth Military Medical University
Locations (1):
- Dingxin, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Merheb J, Van Assche N, Coucke W, Jacobs R, Naert I, Quirynen M. Relationship between cortical bone thickness or computerized tomography-derived bone density values and implant stability. Clin Oral Implants Res. 2010 Jun;21(6):612-7. doi: 10.1111/j.1600-0501.2009.01880.x. PMID 20666788
- [Result] Goodacre CJ, Bernal G, Rungcharassaeng K, Kan JY. Clinical complications with implants and implant prostheses. J Prosthet Dent. 2003 Aug;90(2):121-32. doi: 10.1016/S0022-3913(03)00212-9. PMID 12886205
- [Result] Fugazzotto PA. Success and failure rates of osseointegrated implants in function in regenerated bone for 72 to 133 months. Int J Oral Maxillofac Implants. 2005 Jan-Feb;20(1):77-83. PMID 15747677
- [Result] Atsumi M, Park SH, Wang HL. Methods used to assess implant stability: current status. Int J Oral Maxillofac Implants. 2007 Sep-Oct;22(5):743-54. PMID 17974108
- [Result] Javed F, Romanos GE. The role of primary stability for successful immediate loading of dental implants. A literature review. J Dent. 2010 Aug;38(8):612-20. doi: 10.1016/j.jdent.2010.05.013. Epub 2010 Jun 11. PMID 20546821
- [Result] Herrmann I, Lekholm U, Holm S, Kultje C. Evaluation of patient and implant characteristics as potential prognostic factors for oral implant failures. Int J Oral Maxillofac Implants. 2005 Mar-Apr;20(2):220-30. PMID 15839115
- [Result] Turkyilmaz I, Tozum TF, Tumer C, Ozbek EN. Assessment of correlation between computerized tomography values of the bone, and maximum torque and resonance frequency values at dental implant placement. J Oral Rehabil. 2006 Dec;33(12):881-8. doi: 10.1111/j.1365-2842.2006.01692.x. PMID 17168930
- [Result] Aksoy U, Eratalay K, Tozum TF. The possible association among bone density values, resonance frequency measurements, tactile sense, and histomorphometric evaluations of dental implant osteotomy sites: a preliminary study. Implant Dent. 2009 Aug;18(4):316-25. doi: 10.1097/ID.0b013e31819ecc12. PMID 19667820
- [Result] Farre-Pages N, Auge-Castro ML, Alaejos-Algarra F, Mareque-Bueno J, Ferres-Padro E, Hernandez-Alfaro F. Relation between bone density and primary implant stability. Med Oral Patol Oral Cir Bucal. 2011 Jan 1;16(1):e62-7. doi: 10.4317/medoral.16.e62. PMID 20711163
- [Result] Monje A, Suarez F, Garaicoa CA, Monje F, Galindo-Moreno P, Garcia-Nogales A, Wang HL. Effect of location on primary stability and healing of dental implants. Implant Dent. 2014 Feb;23(1):69-73. doi: 10.1097/ID.0000000000000019. PMID 24384740
- [Result] Turkyilmaz I, Tumer C, Ozbek EN, Tozum TF. Relations between the bone density values from computerized tomography, and implant stability parameters: a clinical study of 230 regular platform implants. J Clin Periodontol. 2007 Aug;34(8):716-22. doi: 10.1111/j.1600-051X.2007.01112.x. PMID 17635248
- [Result] Hong J, Lim YJ, Park SO. Quantitative biomechanical analysis of the influence of the cortical bone and implant length on primary stability. Clin Oral Implants Res. 2012 Oct;23(10):1193-7. doi: 10.1111/j.1600-0501.2011.02285.x. Epub 2011 Sep 29. PMID 22092387
- [Result] Calvo-Guirado JL, Lopez-Lopez PJ, Perez-Albacete Martinez C, Javed F, Granero-Marin JM, Mate Sanchez de Val JE, Ramirez Fernandez MP. Peri-implant bone loss clinical and radiographic evaluation around rough neck and microthread implants: a 5-year study. Clin Oral Implants Res. 2018 Jun;29(6):635-643. doi: 10.1111/clr.12775. Epub 2016 Jan 7. PMID 26744262